CLINICAL TRIAL: NCT02548312
Title: Randomised Controlled Trial to Measure the Effect of Different Financial Competing Interest Statements on Readers' Perceptions of Clinical Educational Articles
Brief Title: The Effect of Different Financial Competing Interest Statements on Readers' Perceptions of Clinical Educational Articles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The BMJ (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COI-RCT
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Readers' perceptions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Review 1- competing interest statement 1 (Experimental): Variations of financial competing interest statements. There will be a statement that the authors have no competing interests.
  Interventions: Other: Variations of financial competing interest statements
- Review 1- competing interest statement 2 (Experimental): Variations of financial competing interest statements.
  Interventions: Other: Variations of financial competing interest statements
- Review 1- competing interest statement 3 (Experimental): Variations of financial competing interest statements.
  Interventions: Other: Variations of financial competing interest statements
- Review 1- competing interest statement 4 (Experimental): Variations of financial competing interest statements.
  Interventions: Other: Variations of financial competing interest statements
- Review 2- competing interest statement 1 (Experimental): Variations of financial competing interest statements. There will be a statement that the authors have no competing interests.
  Interventions: Other: Variations of financial competing interest statements
- Review 2- competing interest statement 2 (Experimental): Variations of financial competing interest statements.
  Interventions: Other: Variations of financial competing interest statements
- Review 2- competing interest statement 3 (Experimental): Variations of financial competing interest statements.
  Interventions: Other: Variations of financial competing interest statements
- Review 2- competing interest statement 4 (Experimental): Variations of financial competing interest statements.
  Interventions: Other: Variations of financial competing interest statements

INTERVENTIONS:
Other: Variations of financial competing interest statements — Participants will be randomised to receive 1 of 2 review articles on different topics. For each review there will be 4 groups. Each of the 4 groups will receive an identical version of the review article with the exception of the competing interest statement which will vary depending on group assignment.

SUMMARY:
Financial ties with industry are common among doctors, academics and institutions. This trial aims to investigate the influence of different types of industry-linked activities on readers' perceptions of clinical reviews. Two clinical reviews have been selected on medical topics and study participants (practicing doctors) will be sent one review each. The reviews will be identical except for the inclusion of one of four different permutations of competing interest statements. Participants will be asked to rate the one review they are sent based on the study outcomes (confidence, interest, importance and likeliness to change practice). The study focus is on educational articles as these are intended to guide patient care and convey the authors' interpretation of selected data.

ELIGIBILITY:
Inclusion Criteria:

* Practising doctors in the UK who are members of the British Medical Association (BMA) and receive The BMJ will be included.

Exclusion Criteria:

* BMA members who have opted out of receiving a free copy of The BMJ, public health doctors, consultant oral/dental surgeons, consultants in private practice, retired doctors and student members will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1065 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Schroter, PhD, Principal Investigator — The BMJ

REFERENCES:
- [Derived] Schroter S, Pakpoor J, Morris J, Chew M, Godlee F. Effect of different financial competing interest statements on readers' perceptions of clinical educational articles: a randomised controlled trial. BMJ Open. 2019 Feb 19;9(2):e025029. doi: 10.1136/bmjopen-2018-025029. PMID 30782923
- [Derived] Schroter S, Pakpoor J, Morris J, Chew M, Godlee F. Effect of different financial competing interest statements on readers' perceptions of clinical educational articles: study protocol for a randomised controlled trial. BMJ Open. 2016 Jun 10;6(6):e012677. doi: 10.1136/bmjopen-2016-012677. PMID 27288389

RESULTS

PARTICIPANT FLOW:
Groups:
- Dyspepsia Review- Competing Interest Statement 1; Gout Review- Competing Interest Statement 1: Honoraria & Travel:
  We have read and understood the BMJ policy on declaration of interests and declare the following: DF is funded by a NIH clinician scientist award; SN receives no specific funding; JB has received honoraria and travel expenses from Jenka Pharmaceuticals for lecturing at a conference.
- Gout Review- Competing Interest Statement 2: Advisory board & consultancies:
  We have read and understood the BMJ policy on declaration of interests and declare the following: DF is funded by a NIH clinician scientist award; SN receives no specific funding; JB has received fees from Jenka Pharmaceuticals for consultancies and being an advisory board member.
- Dyspepsia Review- Competing Interest Statement 3; Gout Review- Competing Interest Statement 3: Research funding:
  We have read and understood the BMJ policy on declaration of interests and declare the following: DF is funded by a NIH clinician scientist award; SN receives no specific funding; JB has received research funding from Jenka Pharmaceuticals
- Dyspepsia Review- Competing Interest Statement 4; Gout Review- Competing Interest Statement 4: None:
  We have read and understood the BMJ policy on declaration of interests and declare the following: DF is funded by a NIH clinician scientist award; SN receives no specific funding; JB has no competing interests.
- Dyspepsia Review- Competing Interest Statement 2: Advisory board & consultancies.
  We have read and understood the BMJ policy on declaration of interests and declare the following: DF is funded by a NIH clinician scientist award; SN receives no specific funding; JB has received fees from Jenka Pharmaceuticals for consultancies and being an advisory board member.
Period: Overall Study
Arm/Group | Dyspepsia Review- Competing Interest Statement 1 | Gout Review- Competing Interest Statement 2 | Dyspepsia Review- Competing Interest Statement 3 | Dyspepsia Review- Competing Interest Statement 4 | Gout Review- Competing Interest Statement 1 | Dyspepsia Review- Competing Interest Statement 2 | Gout Review- Competing Interest Statement 3 | Gout Review- Competing Interest Statement 4
Started | 133 | 133 | 134 | 133 | 133 | 133 | 133 | 133
Completed | 100 | 90 | 96 | 87 | 99 | 93 | 93 | 91
Not Completed | 33 | 43 | 38 | 46 | 34 | 40 | 40 | 42

BASELINE CHARACTERISTICS:
Groups:
- Dyapepsia Review- Competing Interest Statement 2: Advisory board & consultancies.
  We have read and understood the BMJ policy on declaration of interests and declare the following: DF is funded by a NIH clinician scientist award; SN receives no specific funding; JB has received fees from Jenka Pharmaceuticals for consultancies and being an advisory board member.
- Total: Total of all reporting groups
Arm/Group | Dyspepsia Review- Competing Interest Statement 1 | Gout Review- Competing Interest Statement 2 | Dyspepsia Review- Competing Interest Statement 3 | Dyspepsia Review- Competing Interest Statement 4 | Gout Review- Competing Interest Statement 1 | Dyapepsia Review- Competing Interest Statement 2 | Gout Review- Competing Interest Statement 3 | Gout Review- Competing Interest Statement 4 | Total
Number analyzed (Participants) | 100 | 90 | 96 | 87 | 99 | 93 | 93 | 91 | 749
Age, Continuous [Mean (Full Range); unit: years] | 43.5 [23 to 79] | 45.5 [24 to 72] | 44.7 [25 to 75] | 42.8 [24 to 67] | 44.9 [25 to 75] | 42.9 [24 to 76] | 42.8 [24 to 67] | 42.9 [24 to 76] | 44 [23 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 46 | 55 | 45 | 53 | 51 | 51 | 51 | 404
  Male | 48 | 44 | 41 | 42 | 46 | 42 | 42 | 40 | 345
Region of Enrollment [Number; unit: participants]
  United Kingdom | 100 | 90 | 96 | 87 | 99 | 93 | 93 | 91 | 749
Type of doctor [Count of Participants; unit: Participants]
  Consultant | 31 | 33 | 35 | 33 | 37 | 31 | 34 | 30 | 264
  General practice | 36 | 34 | 35 | 29 | 33 | 34 | 33 | 29 | 263
  Junior doctor | 33 | 23 | 26 | 25 | 29 | 28 | 26 | 32 | 222

OUTCOME MEASURES:

1. Primary Outcome: The Readers' Level of Confidence in the Conclusions Drawn in the Article.
Description: Measured on a single-item 10-point Likert scale from (1) "not at all confident" to (10) "extremely confident". Higher scores indicate more confidence. Min score = 0, max score =10.
Time Frame: Outcome measure will be assessed only at the time of the intervention (0 weeks). Readers will be asked to complete the study questionnaire immediately after reading the review article.
Population: One participant in the Group 'Gout review- competing interest statement 2', one in 'Dyspepsia review- competing interest statement 2', one in 'Dyspepsia- statement 3', and one in 'Gout- statement 4' did not respond to the question related to the primary outcome. Hence, for this outcome the numbers analyzed= 89, 92, 95 and 90, respectively.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dyspepsia Review- Competing Interest Statement 1 | Gout Review- Competing Interest Statement 2 | Dyspepsia Review- Competing Interest Statement 3 | Dyspepsia Review- Competing Interest Statement 4 | Gout Review- Competing Interest Statement 1 | Dyspepsia Review- Competing Interest Statement 2 | Gout Review- Competing Interest Statement 3 | Gout Review- Competing Interest Statement 4
Number analyzed (Participants) | 100 | 89 | 95 | 87 | 99 | 92 | 93 | 90
score on a scale | 6.2 [5.8 to 6.6] | 7.0 [6.7 to 7.4] | 6.1 [5.7 to 6.5] | 6.4 [6.0 to 6.8] | 7.1 [6.8 to 7.5] | 6.2 [5.8 to 6.6] | 7.4 [7.1 to 7.8] | 7.4 [7.0 to 7.8]

2. Secondary Outcome: Importance of the Article.
Description: Measured on a single-item 10-point Likert scale from (1) "not at all important" to (10) "extremely important". Higher scores indicate more importance. Min score = 0, max score =10.
  Readers will be asked to complete the study questionnaire immediately after reading the review article.
Time Frame: Outcome measure will be assessed only at the time of the intervention (0 weeks)
Population: One participant in the Group 'Gout review- competing interest statement 4' and one participant in 'Dyspepasia review- competing interest statement 3' did not respond to the question related to this outcome. Hence, for this outcome the numbers analyzed= 90 and 95 respectively (n=91 and n=96 in the participant flow chart).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dyspepsia Review- Competing Interest Statement 1 | Gout Review- Competing Interest Statement 2 | Dyspepsia Review- Competing Interest Statement 3 | Dyspepsia Review- Competing Interest Statement 4 | Gout Review- Competing Interest Statement 1 | Dyspepsia Review- Competing Interest Statement 2 | Gout Review- Competing Interest Statement 3 | Gout Review- Competing Interest Statement 4
Number analyzed (Participants) | 100 | 90 | 95 | 87 | 99 | 93 | 93 | 90
score on a scale | 6.3 [6.0 to 6.7] | 6.4 [6.1 to 6.8] | 6.3 [5.9 to 6.7] | 6.3 [5.9 to 6.7] | 6.9 [6.6 to 7.3] | 6.5 [6.2 to 6.9] | 6.7 [6.4 to 7.1] | 7.0 [6.6 to 7.4]

3. Secondary Outcome: Interest in the Article.
Description: Measured on a single-item 10-point Likert scale from (1) "not at all interesting" to (10) "extremely interesting". Higher scores indicate more interest. Min score = 0, max score =10.
  Readers will be asked to complete the study questionnaire immediately after reading the review article.
Time Frame: Outcome measure will be assessed only at the time of the intervention (0 weeks)
Population: One participant in the Group 'Dyspepsia review- competing interest statement 2', 'Dyspepsia review- statement 3', 'Gout review- statement 4' did not respond to the question related to this outcome. Hence, for this outcome the numbers analyzed= 92, 90 and 95 respectively (however n=93, 91 and 96 in participant flowchart).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dyspepsia Review- Competing Interest Statement 1 | Gout Review- Competing Interest Statement 2 | Dyspepsia Review- Competing Interest Statement 3 | Dyspepsia Review- Competing Interest Statement 4 | Gout Review- Competing Interest Statement 1 | Dyspepsia Review- Competing Interest Statement 2 | Gout Review- Competing Interest Statement 3 | Gout Review- Competing Interest Statement 4
Number analyzed (Participants) | 100 | 90 | 95 | 87 | 99 | 92 | 93 | 90
score on a scale | 5.9 [5.5 to 6.3] | 6.2 [5.9 to 6.6] | 5.8 [5.4 to 6.2] | 5.8 [5.4 to 6.2] | 6.7 [6.5 to 7.0] | 6.0 [5.6 to 6.4] | 6.5 [6.2 to 6.9] | 7.0 [6.7 to 7.4]

4. Secondary Outcome: Number of Participants Who Are Extremely Likely to Change Practice on the Basis of the Article (Scored a "10"), for Those Currently Treating the Relevant Condition
Description: Measured on a single-item 10-point Likert scale from (1) "not at all likely" to (10) "extremely likely". Higher scores indicate more likely to change practice. Min score = 1, max score =10.
  Readers asked to complete the study questionnaire immediately after reading the review article.
Time Frame: Outcome measure will be assessed only at the time of the intervention (0 weeks)
Population: Analysis only includes subset that indicated they currently treat gout/dyspepsia and own practice differed from recommendations given in the review.
Measure: Count of Participants; unit: Participants
Arm/Group | Dyspepsia Review- Competing Interest Statement 1 | Gout Review- Competing Interest Statement 2 | Dyspepsia Review- Competing Interest Statement 3 | Dyspepsia Review- Competing Interest Statement 4 | Gout Review- Competing Interest Statement 1 | Dyspepsia Review- Competing Interest Statement 2 | Gout Review- Competing Interest Statement 3 | Gout Review- Competing Interest Statement 4
Number analyzed (Participants) | 20 | 17 | 29 | 12 | 16 | 19 | 11 | 15
Participants | 0 | 4 | 2 | 1 | 1 | 2 | 2 | 3

ADVERSE EVENTS:
Arm/Group | Dyspepsia Review- Competing Interest Statement 1 | Gout Review- Competing Interest Statement 2 | Dyspepsia Review- Competing Interest Statement 3 | Dyspepsia Review- Competing Interest Statement 4 | Gout Review- Competing Interest Statement 1 | Dyspepsia Review- Competing Interest Statement 2 | Gout Review- Competing Interest Statement 3 | Gout Review- Competing Interest Statement 4
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/90 | 0/96 | 0/87 | 0/99 | 0/93 | 0/93 | 0/91
Other Adverse Events (participants affected / at risk) | 0/100 | 0/90 | 0/96 | 0/87 | 0/99 | 0/93 | 0/93 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No